CLINICAL TRIAL: NCT06031506
Title: Management of Severely Atrophied Maxillary Ridge Using Quad Zygomatic Implants to Support Immediately Loaded Hybrid Prosthesis.One Year Evaluation of Occlusal Contact and Ridge Resorption
Brief Title: Management of Severely Atrophied Maxillary Ridge Using Quad Zygomatic Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M03071221
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: All patients will receive conventional maxillary and mandibular complete dentures The implant size will be selected for each area according to the available bone length and width as measured by CBCT radiograph.
  All implants will be surgically installed guided by steriolethognathic stents
  - Multi-unit abutments will be connected to implants and will be immedietly loaded by fixed full arch screw retained provisional acrylic restoration.
  Final prosthesis will be delivered 6-8 months later
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- quad zygomatic hybrid maxillary prosthesis (Experimental): All patients will be rehabilitated with immediate loaded hybrid prosthesis supported by 4 zygomatic implants.
  Interventions: Device: Implant supported hybrid maxillary prosthesis

INTERVENTIONS:
Device: Implant supported hybrid maxillary prosthesis — All patients will receive immediately loaded hybrid prosthesis supported by 4 zygomatic implants.

SUMMARY:
This clinical study will aim to compare and evaluate zygomatic implant stability, occlusal contact, and bone level changes around dental implants

DETAILED DESCRIPTION:
The aim of this study will be to compare and evaluate zygomatic implant stability, occlusal contact, and bone level changes around dental implants and that of the atrophied maxilla rehabilitated with immediate loaded hyprid prosthesis supported by 4 zygomatic implants.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have healthy healed residual alveolar ridges, Angle's class I maxillomandibular relations, available maxillary restorative space. This will be verified by tentative jaw relation records.

Exclusion Criteria:

* All detrimental bad habits like smoking, TMJ clicking or TMJ dysfunction will be excluded.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | one year
  The patient satisfaction will be evaluated using the visual analog scale (VAS) questionnaire at base line, 6, and 12 months later
marginal implant bone loss | one year
  The implant marginal bone height changes will be measured radiographically at base line, 6, and 12 months later

SECONDARY OUTCOMES:
posterior area index | one year
  the area index of the anterior and posterior maxillary ridge will be measured radiographically at base line, 6, and 12 months later

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No